CLINICAL TRIAL: NCT00771992
Title: Ex Vivo Effect of Surfactant Protein D on Pulmonary Immune Cells Derived From Bronchoalveolar Lavage After Segmental Allergen Challenge in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Prof. Dr. Jens Hohlfeld, Fraunhofer ITEM
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08/09 ZAP-SFB
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Asthma
Keywords: Asthma GINA 1
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy with segmental allergen challenge

SUMMARY:
The effect of surfactant protein D under native and altered conditions will be investigated in immune cells that are derived from bronchoalveolar lavage in patients with allergic asthma following segmental allergen challenge. The goal of this study is to elucidate the pro- versus anti-inflammatory function of SP-D molecules and to identify motifs of SP-D that have treatment potential in allergic asthma.

DETAILED DESCRIPTION:
Following a baseline BAL, allergen (3×) and saline (1×) will be instilled into four different lung segments during a first bronchoscopy. After 24 hours during a second bronchoscopy BAL will be collected in these challenged segments to harvest invaded cells for in-vitro experimentation. In addition, bronchial biopsies and epithelial brushes will be taken to assess the degree of local inflammation in bronchial mucosa and to study the activation of airway epithelium following allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Physician diagnosis of mild asthma according to GINA guidelines (7)
* age 18-55 years
* Nonsmokers with a history of less than 1 packyear having been nonsmokers for at least the last five years
* FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70 %
* Positive skin prick test for grass mix or D. pteronyssinus at or within 12 months prior to the screening visit
* Positive response to inhaled methacholine (≤ 8 mg/mL)
* Positive response to an incremental inhaled allergen challenge with house dust mite allergen or grass pollen allergen
* Women will be considered for inclusion if they are:
* not pregnant, as confirmed by pregnancy test, and not nursing
* of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit)
* of childbearing potential and using a highly effective method of contraception during the entire study (vasectomized partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the study until at least 72 hours after the end of the study -, implants, injectables, combined oral contraceptives, hormonal IUDs, or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap)
* Available to complete all study measurements

Exclusion Criteria:

* History of upper or lower respiratory tract infection four weeks prior to the informed consent visit
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease, or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Clinically significant pathological findings in safety laboratory tests
* Regular intake of any medication other than short acting inhaled beta agonists, paracetamol for pain relief, birth control medication, hormonal replacement therapy, dietary and vitamin supplements
* Specific Immunotherapy (SIT) within two years prior to the study
* Use of anti-inflammatory medication including systemic or inhaled corticosteroid within the last four weeks
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Suspected hypersensitivity to any ingredients of the medication in line with bronchoscopy (bronchodilators, sedatives and local anesthetics)
* Conditions or factors, which would make the subject unlikely to be able to undergo bronchoscopy or incremental allergen challenge
* History of drug or alcohol abuse
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* Participation in a clinical trial 30 days prior to enrolment
* Segmental allergen challenge three months prior to treatment
* Risk of non-compliance with study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
change of numbers of matured dendritic cells in vitro in the absence and presence of surfactant protein D. | 24 h post allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

REFERENCES:
- See also: Related Info — http://www.atemwegsforschung.de